CLINICAL TRIAL: NCT03124329
Title: An Open Prospective Randomized Controlled Clinical Trial to Examine the Efficacy of Methods to Treat Multiple Gingival Recession Defects
Brief Title: Efficacy of Methods to Treat Multiple Gingival Recession Defects
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI has left the organization
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Neema Bakhshalian, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-16-00661
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2019-06

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Coronally Advanced Flap (Experimental)
  Interventions: Procedure: Coronally Advanced Flap
- Vestibular Incision Subperiosteal Tunnel Access (VISTA) (Experimental)
  Interventions: Biological: Vestibular Incision Subperiosteal Tunnel Access (VISTA)
- Intrasulcular tunneling (Experimental)
  Interventions: Procedure: Intrasulcular Tunneling
- VISTA + Leukocyte-Platelet Rich Fibrin (Experimental)
  Interventions: Biological: Vestibular Incision Subperiosteal Tunnel Access (VISTA); Device: Leukocyte-Platelet Rich Fibrin (L-PRF)

INTERVENTIONS:
Procedure: Coronally Advanced Flap — Coronally advanced flap will be performed. Briefly, sulcular incisions will be made. Oblique incisions will be made on each papilla requiring root coverage. In the region coronal to the mucogingival junction (MGJ), mucoperiosteal flap will be elevated. Apical to the MGJ, sharp dissection will be performed to the periosteum allowing split-thickness flap elevation to be performed. Epithelium is removed from the papillae adjacent to the recession and the flap is coronally positioned and stabilized with interproximal sutures and apico-coronal interrupted sutures to close the vertical releasing incisions.
  Arms: Coronally Advanced Flap
Procedure: Intrasulcular Tunneling — Initial sulcular incisions are made and small, contoured blades and mini curettes are used to create the recipient pouches and tunnels. The tunnel will be subperiosteal in location. The incision is extended to one adjacent tooth both mesially and distally. This incision maintains the full height and thickness of the gingival component and enables access beneath the buccal gingiva. The connective tissue beyond the mucogingival line will be dissected and free the buccal flap from its insertions to the bone around each tooth. Muscle fibers and any remaining collagen fibers on the inner aspect of the flap, which prevent the buccal gingiva from being moved coronally, are cut. The papillae are kept intact and undermined to maintain their integrity and carefully released from the underlying bone, which allows the coronal positioning of the papillae. An envelope, full-thickness pouch, and tunnel are created and extended apically beyond the mucogingival line by blunt dissection
  Arms: Intrasulcular tunneling
Biological: Vestibular Incision Subperiosteal Tunnel Access (VISTA) — The VISTA approach begins with a Vestibular Incision Subperiosteal Tunnel Access. Through this incision a subperiosteal tunnel is created, exposing the facial osseous plate and root dehiscence. This tunnel will be extended at least one or two teeth beyond the teeth requiring root coverage to mobilize gingival margins and facilitate coronal repositioning. Additionally, the subperiosteal tunnel is extended interproximally under each papilla as far as the embrasure space permits, without making any surface incisions through the papilla. The mucogingival complex is then advanced coronally and stabilized in the new position with the coronally anchored suturing technique, which entails placing a horizontal mattress suture apical to the gingival margin of each tooth. The suture is tied to position the knot at the midcoronal point of the facial aspect of each tooth, which is secured with help of composite resin to prevent apical relapse of the gingival margin during initial stages of healing.
  Arms: VISTA + Leukocyte-Platelet Rich Fibrin; Vestibular Incision Subperiosteal Tunnel Access (VISTA)
Device: Leukocyte-Platelet Rich Fibrin (L-PRF) — Immediately prior to surgery, 72 mL of blood should be drawn from each patient by venipuncture of the antecubital vein and collected in a sterile glass test tube without any anticoagulant. Tubes should be centrifuged at 2,700 rpm for 12 minutes within 2 minutes after blood draw. For individuals on anti-coagulant therapy or supplements to interfere with coagulation, centrifugation will be for 18 minute. After centrifugation, each L-PRF clot will be separated from the portion of red blood cells (red thrombus), obtaining a fibrin clot with a red small portion in order to include the "buffy" coat richer in leucocytes. The L-PRF clot is condensed and modeled on a sterile surgical plate. L-PRF will be used within 60 minutes after the preparation.
  Arms: VISTA + Leukocyte-Platelet Rich Fibrin

SUMMARY:
Rationale: Treatment of gingival recession defects requires coronal advancement of the gingival margin due to patient esthetic demand, tooth sensitivity and improvement of tooth prognosis, which can be accomplished either through a flap procedure or through a tunnel. It will be desirable to determine the efficacy of Vestibular Incision Subperiosteal Tunnel Access (VISTA) to Coronally Advanced Flap (CAF) procedure and intrasulcular tunneling.

Another aspect of the study is to determine whether autologous concentrate of platelets and leukocytes (leukocyte-platelet-rich fibrin; L-PRF) has equivalent efficacy to connective tissue autologous graft harvested from the palate.

The overall objective of this study is to evaluate the effectiveness of therapeutic modalities for the treatment of multiple gingival recession defects.

The study is designed as a prospective, randomized controlled clinical trial. Four groups will be compared:

Group 1: Coronally Advanced Flap (CAF) Group 2: VISTA Group 3: Intrasulcular tunneling (IST) Group 4: VISTA + L-PRF

Each of the groups will be treated without any graft material in order to examine the efficacy of coronal advancement and periodontal root coverage without the confounding variable of graft material. These techniques don't require any additional graft if there is adequate amount of keratinized gingiva

The study population will be patients who present to Advanced Graduate Program in Periodontology at the University of Southern California, USA, and are deemed to require treatment of multiple gingival recession defects. A total sample of 100 participants (23 participants per group) will provide a two sided test of means with 80% power at alpha of 0.05. The calculation was carried out using PASS Version 12 (Hintze, J. (2014). NCSS, LLC. Kaysville, Utah.)

The study duration will be 1 year. Follow-up visits after the surgery will occur after 3 days , 7 days and at weeks 3, 6, 12, 24, 36 and 52. These follow up visits consistent with standard of care follow up for gingival recession treatment and there will be no additional costs to the participant.

The Primary Outcome variable is complete root coverage; the Secondary Outcome Variables are clinical attachment level (CAL) gain, changes in gingival thickness and volume and the Tertiary Outcomes are aesthetic outcomes, postoperative pain and Patient satisfaction survey

ELIGIBILITY:
Inclusion Criteria:

* Male and female individuals between ages of 18 to 70 years old
* Multiple contiguous gingival recession defects on a minimum of two adjacent teeth, exhibiting 3mm or more recession on at least one of those teeth
* No prior surgical treatment in the sites planned for therapy
* Minimum of 2 mm of keratinized gingiva
* Absence of cervical restorations extending to the CEJ
* Miller class 1, 2 and 3 recession defects will be included
* Availability to undergo treatment and return for follow up visits at specified post-operative intervals

Exclusion Criteria:

* Molar teeth
* Milller Class 4 recession defects
* Pregnancy (Self-reported)
* Smoking
* Uncontrolled local or systemic diseases that affects wound healing (diabetes, autoimmune or inflammatory disorders)
* Past history of systemic steroid use over 2 weeks within the last 2 years
* Poor oral hygiene on a non-compliant individual
* Ibuprofen Allergy/interlerance
* Anticoagulant therapy (e.g. Warfarin, Plavix, etc.), will not be automatic exclusion but patients will be required to have INR test performed and have values between 2.0 to 3. Physician consultation will be requested to determine whether anticoagulant therapy can be discontinued for 3 days prior to surgery.
* Objection to blood draw or application of blood products
* Students and staff from USC Ostrow school of Dentistry will not be recruited for this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Complete root coverage | 12 months
  Complete coverage of the recession defect following surgery. It will be a binary outcome (Yes or No)

SECONDARY OUTCOMES:
Clinical Attachment Level gain | 12 months
  Gain of clinical attachment defined by the distance between the cement-enamel junction to the depth of the periodontal pocket around the teeth measured in mm by a periodontal probe
% root coverage | 12 months
  Percentage of the denuded root surface which is covered following the procedure
Gingival Thickness Gain | 12 months
  Thickness of the gingival following the procedure
Gingival Volume Gain | 12 months
  The gingival volume gain following the procedure

OTHER OUTCOMES:
Patient-reported outcomes | 3 days
  Includes: pain experienced within the mouth as a whole, pain experienced while drinking beverages, pain experienced while chewing, pain experienced in the morning, Pain experienced throughout the day, Pain experienced at night, Edema experienced after the surgery all measure with the use of a Visual Analogue Scale
objective esthetic assessment | 6 months
  This score evaluates five variables: level of the gingival margin, marginal tissue contour, soft tissue texture, mucogingival junction alignment, and gingival color. Because complete root coverage is the primary treatment goal, and the other variables were considered secondary, the value assigned for root coverage is 60% of the total score, whereas 40% is assigned to the other four variables.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The intra-oral clinical photography, CBCT scans, study models and clinical data will be shared with other investigators for data analysis.